CLINICAL TRIAL: NCT00896779
Title: Lucentis in Advanced Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Steven R. Sanislo (Other)
Collaborators: Genentech, Inc. (Industry); California Pacific Medical Center (Other); Pacific Eye Associates (Other)
Responsible Party: Sponsor-Investigator, Steven R. Sanislo, MD/PI, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-04202009-2338
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ranibizumab Group 1 (Other): Group 1: 3 monthly injections of 0.5mg then prn
  Interventions: Drug: ranibizumab
- ranibizumab Group 2 (Other): Group 2: 6 monthly injections of 0.5 mg then prn
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — Group 1 - 0.5mg intravitreal injection every month for 3 months then as needed for 12 months
  Group 2 -0.5mg intravitreal injection every month for 6 months then as needed for 12 months
  Other Names: Lucentis

SUMMARY:
Patients with low vision (visual acuity 20/400 or worse) were excluded from the large Phase III ranibizumab clinical trials. It is not known if treatment with ranibizumab results in improved visual function in such patients.Since ranibizumab has been shown to be the most effective therapy for exudative macular degeneration we propose to treat all patients in this study with monthly ranibizumab intravitreal injections.

Patients will be assigned to one of two groups by the flip of a coin. Group #1 for "heads" and Group #2 for "tails".

Group #1 patients will be treated for 3 monthly injections of 0.5 mg of ranibizumab and then as needed therapy.

Group #2 will be treated with 6 monthly injections of 0.5 mg of ranibizumab and then as needed therapy.

DETAILED DESCRIPTION:
The duration of the study is up to 13 months. This includes up to 30 days during which tests will be performed before treatment. Only one eye will be chosen for the study. Patients can receive up to 12 injections of ranibizumab during this study (the first dose[s], plus additional doses [re treatment as often as every 22 days] if the doctor determines that additional doses are required).

In addition to study drug injections. Several eye examinations and procedures will be performed to evaluate response to treatment. These include: visual acuity testing (eye chart), contrast sensitivity testing, reading speed testing, measurement of time to complete typical daily activities, measurement of the thickness of the central retina, measurement of your central visual field.

On the screening visit and two more times during the study fluorescein angiography will be performed.

The screening tests included the following:

* A review of your medical history
* A review of any medications you are or have been taking
* Eye examinations, including visual acuity testing (reading letters on an eye chart)
* Blood pressure measurement Woman of childbearing potential must also take a urine pregnancy test during the screening period to rule out pregnancy.

Upon completion of the study at Month 12 and if it were to occur; early termination visit, the following procedures will be performed: vision exam,OCT,microperimetry,FA/Photos,VFQ,reading performance, contrast sensitivity and TIADL.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible if the following criteria are met:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Age > 50 years.
* Low vision AMD patients with a VA of 20/400 or worse.
* Evidence of active exudation as manifested by subretinal or intraretinal fluid on OCT or fresh appearing subretinal hemorrhage on fundus examination.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from this study:

* Pregnancy (positive pregnancy test) or lactation.
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated.
* Participation in another simultaneous medical investigation or trial.
* Concurrent eye disease in the study eye that could compromise visual acuity (e.g., diabetic retinopathy, advanced glaucoma).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Steven R. Sanislo, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - California Pacific Medical Center, San Francisco, California
  - Stanford University School of Medicine, Stanford, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Ranibizumab Group 1: Group 1: 3 monthly injections of raibizumab 0.5mg then injections as needed for 12 months
- Ranibizumab Group 2: Group 1: 6 monthly injections of raibizumab 0.5mg then injections as needed for 12 months
Period: Overall Study
Arm/Group | Ranibizumab Group 1 | Ranibizumab Group 2
Started | 8 | 12
Completed | 8 | 11
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ranibizumab Group 2: Group 2: 6 monthly injecions of 0.5mg then prn
- Total: Total of all reporting groups
Arm/Group | Ranibizumab Group 1 | Ranibizumab Group 2 | Total
Number analyzed (Participants) | 8 | 12 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 8 | 12 | 20
Age, Continuous [Mean (Full Range); unit: years] | 81 [68 to 94] | 84 [71 to 97] | 83 [68 to 97]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 11
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 8 | 12 | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Visual Acuity
Description: Change in vision from baseline measurement at 12 months. Standard ETDRS chart (80 letters) was used to determine visual acuity with test luminance of 45 cd/m ^2 at 8 feet. Number of correctly read letters were reported.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: letters
Groups:
- Ranibizumab Group 2: Group 2: 6 monthly injections of raibizumab 0.5mg then injections as needed for 12 months
Arm/Group | Ranibizumab Group 1 | Ranibizumab Group 2
Number analyzed (Participants) | 8 | 12
letters | 15.0 (14.2) | 5.6 (8.6)
Statistical Analysis 1: Comparison: Ranibizumab Group 1; Test type: Superiority or Other; p = 0.02, t-test, 2 sided
Statistical Analysis 2: Comparison: Ranibizumab Group 2; Test type: Superiority or Other; p = 0.06, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Ranibizumab Group 1 | Ranibizumab Group 2
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/12
Other Adverse Events (participants affected / at risk) | 4/8 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranibizumab Group 1 (N=8) | Ranibizumab Group 2 (N=12)
laceration right leg (Skin and subcutaneous tissue disorders) | 1 | 0
laceration left leg (Skin and subcutaneous tissue disorders) | 1 | 0
Mild pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Seasonal allergies (Immune system disorders) | 1 | 0
Worsening glaucoma - which eye was not specified (Eye disorders) | 1 | 0
visual disturbance - fellow eye (Eye disorders) | 1 | 0
development of choroidal neovascularization - fellow eye (Eye disorders) | 1 | 0
bruised sturnum (Musculoskeletal and connective tissue disorders) | 1 | 0 — Due to auto accident
subconjuctival hemorrhage - treatment eye (Eye disorders) | 1 | 0
intraretinal hemorrhage - treatment eye (Eye disorders) | 1 | 0
vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
intestinal flu (Gastrointestinal disorders) | 1 (2) | 0
rash (Skin and subcutaneous tissue disorders) | 1 | 0
pinched nerve (Nervous system disorders) | 1 | 0
stroke (Nervous system disorders) | 0 | 1
endophthalmitis - fellow eye (Eye disorders) | 0 | 1
cold (Immune system disorders) | 0 | 1
ache left eye - treatment eye (Eye disorders) | 0 | 1 — after injection procedure
corneal abrasion - both eyes (Eye disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Limitations include small number of subjects analyzed and no control group that were untreated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No